CLINICAL TRIAL: NCT02737566
Title: Small Financial Incentives to Promote Smoking Cessation in Safety Net Hospital Patients
Brief Title: Small Financial Incentives to Promote Smoking Cessation
Acronym: Prevail II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6260; R01CA197314 (NIH)
Record Dates: First submitted 2016-04-07; First posted 2016-04-14 (Estimated); Results first posted 2023-04-20 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Financial Incentives; Contingency Management; Vulnerable Populations; Medically Uninsured; Medicaid
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care + Financial Incentives (Experimental): Participants randomized to Standard Care + Financial Incentives for Abstinence will be offered smoking cessation counseling and pharmacotherapy (standard care) and they will have the opportunity to earn small gift cards for biochemically-verified abstinence through 12 weeks post-quit. The amount of the gift cards will escalate each week from the quit date through 4 weeks post-quit with continuous abstinence. Participants who are non-abstinent at any visit may earn incentives for abstinence at the next visit, but the amount will reset to the starting level. Participants may additionally earn an additional gift card for abstinence at the 8 and 12 weeks post-quit visits.
  Interventions: Behavioral: Standard Care + Financial Incentives
- Standard Care (Active Comparator): Participants randomized to Standard Care will be offered weekly smoking cessation counseling and pharmacotherapy.
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Standard Care + Financial Incentives — Tobacco cessation counseling plus pharmacotherapy and financial incentives for quitting.
  Arms: Standard Care + Financial Incentives
Other: Standard Care — Tobacco cessation counseling plus pharmacotherapy.
  Arms: Standard Care

SUMMARY:
The primary objectives of this study are 1) to evaluate the longer-term impact of an adjunctive, low-cost financial incentives intervention (relative to standard care) on smoking abstinence rates among socioeconomically disadvantaged individuals participating in a clinic-based smoking cessation program and 2) to identify treatment mechanisms and contextual factors associated with cessation outcomes among intervention participants using both traditional and ecological momentary assessment approaches. Those randomized to the financial incentives intervention will have the opportunity to earn small gift cards for biochemically-verified abstinence through 12 weeks post-quit. We hypothesize that individuals who are randomly assigned to the adjunctive CM intervention will have significantly higher rates of biochemically-verified abstinence at the 26-week post-quit follow-up than those assigned to Usual Care. In addition, we hypothesize that several factors related to socioeconomic disadvantage will be directly associated with non-abstinence, especially greater stress/adversity, limited psychosocial resources, greater negative affect, greater nicotine dependence, and poorer treatment adherence. The primary study endpoints will include self-reported tobacco use/abstinence, expired carbon monoxide (CO) levels (i.e., the amount of carbon monoxide present in an individual's breath when they breathe out), and saliva cotinine levels at 26 weeks post-quit attempt, though smoking status will be assessed at all visits. Traditional questionnaire measurement and ecological momentary assessment (EMA) will be utilized to measure potential treatment mechanisms including motivation, self-efficacy, and treatment adherence. Other variables including stress/adversity, psychosocial resources, negative affect, nicotine dependence, and treatment adherence will also be assessed.

DETAILED DESCRIPTION:
Individuals (N = 320) will be recruited during their initial visit to the Tobacco Cessation Clinic. Eligible participants (N = 320) will be randomized to: 1) Standard Care, which is counseling and pharmacological treatment (SC; n = 160), or 2) SC + adjunctive financial incentives through 12 weeks post-quit (CM; n = 160). All participants will be followed weekly from 1 week pre-quit through 4 weeks post-quit, and will return for visits at 8, 12, and 26 weeks post-quit. Biochemically verified 7-day point prevalence abstinence will be assessed at all visits, though abstinence at 26 weeks post-quit (longer-term abstinence) will serve as the primary outcome variable. Those randomized to the CM intervention will have the opportunity to earn small gift cards for biochemically-verified abstinence through 12 weeks post-quit. The value of the gift cards will escalate weekly with continuous abstinence from the quit date through 4 weeks post-quit. Additional gift cards for abstinence may be earned at 8 and 12 weeks post-quit. We also hope to gain a better understanding of CM treatment mechanisms and to identify other factors that directly influence cessation via traditional questionnaire and smartphone-based ecological momentary assessment approaches. Smartphone technology allows for "real-time" data collection to more accurately capture important cessation-related variables, and will be used to deliver gain-framed messages to support and strengthen the CM intervention. Participants will complete traditional questionnaire measures on a laptop computer weekly from 1 week pre-quit through 4 weeks post-quit, and at 8, 12, and 26 weeks post-quit. Assessments will be completed by participants either before or after their counseling appointments, for which they will receive reimbursement in the form of gift cards. Participants will also receive a smartphone at the 1 week pre-quit visit and they will be asked to carry it with them at all times through 4 weeks post-quit in order to complete EMAs (5 weeks total). Participants will be prompted to complete EMA assessments 5 times per day (4 random assessments + 1 daily diary) for five consecutive weeks. Participants will be compensated upon the return of the smartphone, based on the percentage of random/daily diary assessments that they completed.

Description of Standard Care. According to the Clinical Practice Guideline, currently recommended components of an intensive tobacco treatment intervention include 1) initial assessment of willingness to participate, 2) the use of multiple types of clinicians (e.g., medical, non-medical), 3) at least 4 treatment sessions, in an individual- or group-counseling format, that are greater than 10 minutes in duration, 4) counseling that includes problem-solving, skills training, and social support components, and 5) and the opportunity to use effective medications to aid in tobacco cessation (e.g., nicotine patch, varenicline). The clinic currently offers all components of standard care. Specifically, individuals who would like to quit smoking are referred (typically via electronic medical record). Patients are scheduled for their initial appointment with a Tobacco Treatment Specialist for an individual counseling session and to discuss pharmacological treatment options. Nicotine replacement therapy is provided during the session, or other medications are prescribed via communication with the patient's physician or by a provider on-site. Those enrolled in the current study will be encouraged to attend at least 5 weekly group sessions to facilitate follow-up and the delivery of study incentives.

Visit 1, Part 1 (Recruitment/Screening). Individuals attending the initial clinic intake session will be provided with a 1-page informational handout with information about the study. After the session, study staff will check in with potential participants regarding their interest. Study staff will review the consent form with interested participants, and they will be screened for eligibility on-site in a private room in the clinic. Participant eligibility for the current study will not influence eligibility for standard treatment through the clinic. The Rapid Estimate of Adult Literacy in Medicine (REALM; see Appendix A) will be administered to ensure that all participants are able to read at ≥ sixth grade level (i.e., required to complete EMA and self-report questionnaires). Expired carbon monoxide (CO) will be measured with a Vitalograph BreathCO carbon monoxide monitor. Participants will be questioned about their 1) insurance status 2) age, 3) current level of smoking, 4) willingness to quit smoking, and 5) willingness/ability to attend 6 weekly sessions (including the first visit). Eligible participants may complete the assessment portion of visit 1.

Visit 1, Part 2 (Pre-Quit Assessment). Participants will complete self-report questionnaires on a laptop computer; and expired CO, weight, and height will be measured in a private room to ensure confidentiality. Participants will be provided with an Android smartphone and instructed regarding the use of the phone (participants may make personal calls) as well as the EMA procedures. Participants will receive 4 random prompts and 1 daily diary prompt (in the morning) during the normal waking hours each day for four consecutive weeks. Participants will be instructed to quit smoking at bedtime or 10:00 pm (whichever occurs first), on the evening prior to their next scheduled counseling session (one week later). Participants will be randomized to Standard Care (SC) or CM using a random numbers table and advised of their group assignment at the conclusion of visit 1. The appropriate schedule of payments (SC or CM) will be discussed with all participants (see Table 1). Visit 1 takes approximately 1 hour to complete, and participants will be scheduled to return for visit 2.

Visit 2 (Quit Day). Participants will complete self-report questionnaires on a laptop computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Visit 2 takes approximately 40 minutes to complete. Participants randomized to the CM treatment will receive an additional payment if they self-report abstinence from smoking since 10 p.m. the prior evening, and their expired is CO level is < 10 ppm (please note that the less stringent cut-off of 10 ppm will be used to verify abstinence at the first visit only, due to the recency of quitting). Participants who do not attend will be contacted by phone to obtain their self-reported smoking status only.

Visit 3 (1 Week Post-Quit). Participants will complete self-report questionnaires on a laptop computer; and expired carbon monoxide (CO) and weight will be measured in a private room to ensure confidentiality. Visit 3 takes approximately 30 minutes to complete. Participants randomized to the CM treatment will receive an additional payment if they self-report continuous abstinence from smoking since the quit day and have an expired CO level of ≤ 6 ppm. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

Visit 4 (2 Weeks Post-Quit). Expired carbon monoxide (CO) and weight will be measured in a private room to ensure confidentiality. The visit 4 assessment takes approximately 5 minutes to complete. Participants randomized to the CM treatment will receive payment if they self-report continuous abstinence from smoking since the quit date and have an expired CO level of ≤ 6 ppm. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

Visit 5 (3 Weeks Post-Quit). Expired carbon monoxide (CO) and weight will be measured in a private room to ensure confidentiality. The visit 5 assessment will take approximately 5 minutes to complete. Participants randomized to the CM treatment will receive payment if they self-report continuous abstinence from smoking since the quit date and have an expired CO level of ≤ 6 ppm. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

Visit 6 (4 Weeks Post-Quit). Participants will complete self-report questionnaires on a laptop computer; and expired CO and weight will be measured in a private room to ensure confidentiality. The visit 6 assessment will take approximately 50 minutes to complete. Upon return of the smartphones, participants will be compensated based on the percentage of completed random assessments. Participants who do not attend will be contacted by phone and/or mail to request that the phone be returned by mail (postage paid envelopes will be sent) or in-person at the next visit. When participants return the phone they will be compensated according to the compensation schedule described above. Participants randomized to the CM treatment will receive an additional payment if they self-report continuous abstinence from smoking since the quit date and have an expired CO level of ≤ 6 ppm. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

Visit 7 (8 Weeks Post-Quit). Participants will complete self-report questionnaires on a laptop computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will receive a payment for completion of the in-person assessments, which will take approximately 30 minutes to complete. Participants randomized to the CM treatment will receive an additional payment if they self-report abstinence from smoking over the past 7 days and have an expired CO level of ≤ 6 ppm. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

Visit 8 (12 Weeks Post-Quit). Participants will complete self-report questionnaires on a laptop computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will receive a payment for completion of the in-person assessments, which will take approximately 30 minutes to complete. Participants randomized to the CM treatment will receive an additional payment if they self-report abstinence from smoking over the past 7 days and have an expired CO level of ≤ 6 ppm. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

Visit 9 (26 Weeks Post-Quit Follow-Up). Participants will complete self-report questionnaires on a laptop computer; and expired CO and weight will be measured in a private room to ensure confidentiality. Participants will receive a payment for completion of the in-person assessments, which will take approximately 40 minutes to complete. Saliva cotinine will also be measured via NicAlert test strips to provide additional evidence of abstinence. Participants who do not attend will be contacted by phone to obtain their self-reported smoking status.

ELIGIBILITY:
Inclusion Criteria:

1. are currently uninsured or receiving Medicaid benefits
2. earn a score ≥ 4 on the REALM indicating > 6th grade English literacy level
3. are willing to quit smoking 7 days from their first visit
4. are ≥ 18 years of age
5. have an expired CO level ≥ 8 ppm suggestive of current smoking
6. are currently smoking ≥ 5 cigarettes per day
7. are willing and able to attend 9 study visits.

Exclusion Criteria:

1. are unwilling to quit smoking 7 days from their first visit
2. have already quit smoking
3. earn a score <4 on the REALM indicating < 7th grade literacy level
4. produce an expired CO level < 8 ppm
5. are currently smoking < 5 cigarettes per day
6. are unwilling or unable to attend study visits
7. are < 18 years of age
8. are not uninsured or receiving Medicaid benefits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang M, Koslovsky MD, Hebert ET, Kendzor DE, Businelle MS, Vannucci M. Bayesian continuous-time hidden Markov models with covariate selection for intensive longitudinal data with measurement error. Psychol Methods. 2023 Aug;28(4):880-894. doi: 10.1037/met0000433. Epub 2021 Dec 20. PMID 34928674
- [Result] Kendzor DE, Businelle MS, Frank-Pearce SG, Waring JJC, Chen S, Hebert ET, Swartz MD, Alexander AC, Sifat MS, Boozary LK, Wetter DW. Financial Incentives for Smoking Cessation Among Socioeconomically Disadvantaged Adults: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2418821. doi: 10.1001/jamanetworkopen.2024.18821. PMID 38954415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care + Financial Incentives | Standard Care
Started | 159 | 161
Completed | 104 | 105
Not Completed | 55 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care + Financial Incentives | Standard Care | Total
Number analyzed (Participants) | 159 | 161 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Missing age for 1 participant.
  years
    number analyzed (Participants) | 158 | 161 | 319
    (all) | 49.0 (11.1) | 48.9 (12.2) | 48.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 96 | 202
  Male | 53 | 65 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 152 | 153 | 305
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 4 | 13
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 36 | 46 | 82
  White | 101 | 99 | 200
  More than one race | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 159 | 161 | 320
Cigarettes Smoked Per Day (pre-quit) [Mean (Standard Deviation); unit: Cigarettes smoked per day] — Population: Missing cigarettes smoked per day for 1 participant.
  Cigarettes smoked per day
    number analyzed (Participants) | 158 | 161 | 319
    (all) | 19.1 (10.2) | 19.2 (10.1) | 19.1 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-verified Smoking Cessation
Description: The primary outcome measure is carbon monoxide (CO)-verified 7-day point prevalence abstinence at 26 weeks post-quit (intent-to-treat; missing=smoking).
Time Frame: 26 weeks post-quit
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care + Financial Incentives | Standard Care
Number analyzed (Participants) | 159 | 161
Participants | 22 | 14

2. Secondary Outcome: Biochemically-verified Smoking Cessation
Description: The secondary outcome measure is Carbon Monoxide (CO)-verified 7-day point prevalence abstinence at 12 weeks post-quit (intent-to-treat; missing=smoking).
Time Frame: 12 weeks post-quit
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care + Financial Incentives | Standard Care
Number analyzed (Participants) | 159 | 161
Participants | 45 | 18

ADVERSE EVENTS:
Time Frame: 27 weeks (1 week pre-quit-date through 26 weeks post-quit-date)
Arm/Group | Standard Care + Financial Incentives | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/161
Other Adverse Events (participants affected / at risk) | 2/159 | 2/161
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Care + Financial Incentives (N=159) | Standard Care (N=161)
Blood in Urine (Renal and urinary disorders) | 0 | 1 — The symptom was not likely related to the study.
Fatigue (Product Issues) | 1 | 0 — Possibly related to varenicline. Participant switched to bupropion.
Dissatisfaction with compensation (Social circumstances) | 1 | 0 — Participant was very dissatisfied with reduced compensation associated with non-compliance (even though this was noted in consent form).
Study smartphone was stolen (Social circumstances) | 0 | 1

LIMITATIONS AND CAVEATS:
Study enrollment occurred from 2017-2021. As a result, a total of 146 (45.6%) of participants received treatment and/or had scheduled study assessments following the onset of the COVID-19 pandemic (in March 2020). The pandemic may have affected smoking cessation outcomes and other study variables, including retention and study follow-up rates through a variety of influences (e.g., institutional restrictions on research, financial, stress/mental health).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT02737566/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT02737566/ICF_001.pdf